CLINICAL TRIAL: NCT03081351
Title: Extended Retroperitoneal Lymphadenectomy and Nerve Plexus Clearance Versus Standard Lymphadenectomy in Pancreaticoduodenectomy for Adenocarcinoma of the Pancreatic Head in a Chinese Population:A Multicenter, Open-label, Randomized Controlled Clinical Trial.
Brief Title: Extended Retroperitoneal Lymphadenectomy and Nerve Plexus Clearance Versus Standard Lymphadenectomy in Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Huashan Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Changhai Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Jiangsu Provincial People's Hospital (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20170305
Record Dates: First submitted 2017-03-05; First posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Pancreaticoduodenectomy
Keywords: Extended retroperitoneal lymphadenectomy, Nerve plexus clearance, Survival benefit

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extended lymphadenectomy and nerve clearance (Experimental): The investigators will implement the pancreaticoduodenectomy using the principle of "Total Peripancreas Excision" to resect the lymph node and nerve plexus. The lymph node include standard 5,6,8a,12b1,12b2,12c,12a-b,14a-b,17a-b and extended 8p,9,12a,12p,14a-d,16a2,16b1 of the abdominal lymph node.
  Interventions: Procedure: extended lymphadenectomy and nerve clearance
- standard lymphadenectomy (Experimental): The investigators will implement the pancreaticoduodenectomy using the standard lymphadenectomy. The lymph node include 5,6,8a,12b1,12b2,12c,12a-b,14a-b,17a-b of the abdominal lymph node.
  Interventions: Procedure: standard lymphadenectomy

INTERVENTIONS:
Procedure: extended lymphadenectomy and nerve clearance — The investigators will implement the pancreaticoduodenectomy using the principle of "Total Peripancreas Excision" to resect the lymph node and nerve plexus. The lymph node include standard 5,6,8a,12b1,12b2,12c,12a-b,14a-b,17a-b and extended 8p,9,12a,12p,14a-d,16a2,16b1 of the abdominal lymph node.
  Arms: extended lymphadenectomy and nerve clearance
Procedure: standard lymphadenectomy — The investigators will implement the pancreaticoduodenectomy using the standard lymphadenectomy. The lymph node include 5,6,8a,12b1,12b2,12c,12a-b,14a-b,17a-b of the abdominal lymph node.
  Arms: standard lymphadenectomy

SUMMARY:
This clinical trial is about the survival benefit of extended lymphadenectomy and nerve clearance versus standard lymphadenectomy in pancreaticoduodenectomy of pancreatic adenocarcinoma，which is a multicenter，prospective，ramdomized clinical trials.

DETAILED DESCRIPTION:
The purpose of this clinical trial is for assessing the survival benefit of extended lymphadenectomy and nerve clearance versus standard lymphadenectomy in pancreaticoduodenectomy of pancreatic adenocarcinoma. And we will focus on the R0 resection using LEEPP(Leeds Pathology Protocol) methods to check whether the tumor is eradicated or not.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years; Karnofsky performance>70; preoperative diagnosis as resectable pancreatic head cancer; patients' relative have signed consent form.

Exclusion Criteria:

* also have severe cardiopulmonary disease, autoimmune disease, chronic renal failure disease; recurrent pancreatic tumor or unresectable tumor; benign pancreatic tumor; also have other malignant tumors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, assessed up to 100 months
  The overall survival of the patients from the time of surgery until the date of pass-away.

SECONDARY OUTCOMES:
Disease free survival | From date of randomization until the date of first documented progression( local recurrence or metastasis), assessed up to 100 months.
  The time of the surgery until the date of the local recurrence or metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jang JY, Kang MJ, Heo JS, Choi SH, Choi DW, Park SJ, Han SS, Yoon DS, Yu HC, Kang KJ, Kim SG, Kim SW. A prospective randomized controlled study comparing outcomes of standard resection and extended resection, including dissection of the nerve plexus and various lymph nodes, in patients with pancreatic head cancer. Ann Surg. 2014 Apr;259(4):656-64. doi: 10.1097/SLA.0000000000000384. PMID 24368638